CLINICAL TRIAL: NCT02021916
Title: Louisville Cooperative Tissue Biorepository of the James Graham Brown Cancer Center Tissue Collection Consent
Brief Title: Louisville Cooperative Tissue Biorepository
Acronym: LCTB
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, Professor, University of Louisville
Other Study IDs: 397.05
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Normal and Abnormal Tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collection of normal or abnormal tissue at the time of surgery from consented subjects. Collection of blood and urine the day of consent or day of surgery.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To provide appropriate collection, storage, and distribution of specimens and medical data to local investigators who have approved IRB protocols for their specific research purposes.

DETAILED DESCRIPTION:
The mission of the Louisville Cooperative Tissue Biorepository is to appropriately collect normal and abnormal tissues that are removed from the human body as a part of standard medical and surgical practice after adequate portions are secured by surgical pathologists to allow for correct diagnoses to be made. The LCTB securely stores appropriately collected human samples for research purposes and appropriately allocates these samples to local investigators for research purposes. The LCTB team appropriately documents all points in the process of obtaining informed consent, collection, storage, and allocation of tissues.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for removal or normal and abnormal tissues as part of standard medical and surgical practice

Exclusion Criteria:

* Patients with known systematic infections including septic patients with bacterial and viral infections, hepatitis, HIV, TB and other defined pathogens will not be included.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery for removal of normal or abnormal tissues that are removed from the human body as part of standard medical and surgical practice at the University of Louisville Hospital, Norton Hospital downtown, Jewish Hospital downtown and Kosair Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 17499 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Collect normal and abnormal tissues that are removed from the human body as a part of standard surgical practice after adequate portions are secured by surgical pathologists to allow for correct diagnoses to be made. | 15 Years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States